CLINICAL TRIAL: NCT06280027
Title: Effect of Midline Discrepancy and Crown Width Disproportion on Perception of Smile Esthetics
Brief Title: Effect of Midline Discrepancy and Crown Width Disporportion on Esthetics
Status: Completed | Type: Observational
Sponsor: Marmara University (Other)
Responsible Party: Sponsor
Other Study IDs: MUDHF_BK1
Record Dates: First submitted 2024-02-20; First posted 2024-02-28 (Actual); Last update posted 2024-02-28 (Actual); Status verified 2024-02

CONDITIONS: Esthetics, Dental
Keywords: Esthetics, Dental; Midline Discrepancy; Crown Width Disproportion
MeSH Terms: interventions — Surveys and Questionnaires

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Cross-Sectional
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (2):
- group1: patients (laypeople) of the university clinic. The inclusion criteria were age ≥18 and ≤70 years.
  Interventions: Other: survey
- group2: restorative dentists and prosthodontists with similar levels of clinical experience (at least 3 years of academic training). The inclusion criteria were age ≥18 and ≤70 years.
  Interventions: Other: survey

INTERVENTIONS:
Other: survey — An online survey was generated to quantitatively evaluate the level of esthetic perception.

SUMMARY:
In the web-based cross-sectional study 180 participants were included. Half of them (n = 90) were patients (laypeople) of the university clinic and the remaining half were restorative dentists and prosthodontists with similar levels of clinical experience (at least 3 years of academic training).

A frontal view full-face portrait image of a 25-year-old female was selected as a model for the study, with a smile exhibiting good dental alignment, a quite good midline position, and tooth size symmetry.

The original image was digitally modified by a single restorative instructor using Photoshop CC (Adobe, USA) software program. The modifications were divided into three parts. The first part was the generation of midline discrepancy at different levels. The midline was digitally moved to the right side of the patient 1 - 4 millimeters, gradually. The midline movement was performed together with the whole maxillary arch.

The second part was the generation of individual crown width disproportions. Accordingly, the mesiodistal width of the left central, lateral, and canine was digitally decreased one by one, gradually, while the width of the symmetrical teeth on the right side was simultaneously increased.

The third part was the generation of distributed crown width disproportions. Accordingly, the total mesiodistal width of the left central, lateral, and canine was equally decreased, gradually, while the total width of the symmetrical teeth on the right side was simultaneously increased.

In total, 15 images were displayed in random order to the participants including the original image. An online survey was generated to quantitatively evaluate the level of esthetic perception. Subsequently, the participants were asked to evaluate the level of smile esthetics of the presented random images, without being informed about the digital manipulations of the images. The participants were even not informed about the original image. They were expected to answer the question "How esthetic do you consider this smile?" The evaluation of each image was performed via a Visual analog scale VAS, ranging from point 0 (extremely not esthetic) to point 100 (extremely esthetic).

DETAILED DESCRIPTION:
The web-based cross-sectional study was designed and conducted in a university clinic between June and December 2023. 180 participants were included in the study. Half of them (n = 90) were patients (laypeople) of the university clinic and the remaining half were restorative dentists and prosthodontists with similar levels of clinical experience (at least 3 years of academic training).

A frontal view full-face portrait image of a 25-year-old female was selected as a model for the study, with a smile exhibiting good dental alignment, a quite good midline position, and tooth size symmetry. A perfectly symmetrical face was not demanded for the model in this study as the human face is considered usually not symmetrical. The frontal smiling image was captured using a DSLR full-frame camera (D750, Nikon, Japan), a macro objective (105 mm VR Nikkor, Nikon), and a dual paraflash/softbox (VL400, Visico, China). The image was saved in RAW data format and named as the original image.

The original image was digitally modified by a single restorative instructor using Photoshop CC (Adobe, USA) software program. The modifications were divided into three parts. The first part was the generation of midline discrepancy at different levels. The midline was digitally moved to the right side of the patient 1 - 4 millimeters, gradually. The midline movement was performed together with the whole maxillary arch. Simultaneously, the maxillary right first molar was gradually darkened to provide a natural-like space at the right buccal corridor.

The second part was the generation of individual crown width disproportions. Accordingly, the mesiodistal width of the left central, lateral, and canine was digitally decreased one by one, gradually, while the width of the symmetrical teeth on the right side was simultaneously increased. Therefore, disproportions of 1 mm and 2 mm were digitally generated for each tooth. For instance, to achieve 1 mm of disproportion on the central incisor, the left central width was decreased by 0.5 mm, while the right central width was increased by 0.5 mm.

The third part was the generation of distributed crown width disproportions. Accordingly, the total mesiodistal width of the left central, lateral, and canine was equally decreased, gradually, while the total width of the symmetrical teeth on the right side was simultaneously increased. Therefore, the distributed disproportions of 1 - 4 mm were digitally generated for the group of teeth. For instance, to achieve 1 mm of distributed disproportion, the total width of the left central, lateral, and canine was decreased by 0.5 mm, and the total width of the anterior teeth on the right side was increased by 0.5 mm. 0.5 mm was shared equally by each tooth. Simultaneously, the maxillary right first molar was gradually darkened to provide a natural-like space at the right buccal corridor.

In total, 15 images were displayed in random order to the participants including the original image. An online survey was generated to quantitatively evaluate the level of esthetic perception. At the beginning of the survey, the participants declared their profession, age, and gender. All the images were presented to the participants on a digitally calibrated monitor (iPad Pro 12.9", Apple Inc., USA) to minimize the standardization limitations. Subsequently, the participants were asked to evaluate the level of smile esthetics of the presented random images, without being informed about the digital manipulations of the images. The participants were even not informed about the original image. They were expected to answer the question "How esthetic do you consider this smile?" The evaluation of each image was performed via a Visual analog scale VAS, ranging from point 0 (extremely not esthetic) to point 100 (extremely esthetic). The participants moved a tab on the visual analog scale to a new position, based on their subjective perception of the presented smile esthetics. The scorings were carried out during midday (10:00 AM-14:00 PM), with standardized artificial lighting conditions and without directly exposing the monitor to the sunlight. The distance between the participant and the screen was consistently 60 cm, which stands for the typical distance between two people during social contact. Each participant could complete the survey once without a time limit and was limited to performing again. A total of 180 participants completed the survey.

ELIGIBILITY:
Inclusion Criteria:

- For Group 1: Patients (laypeople) of the university clinic

* For Group 2:

Restorative dentists and prosthodontists with similar levels of clinical experience (at least 3 years of academic training).

Exclusion Criteria:

* people with mental illness

Ages: 18 Years to 70 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Study Population: Half of them (n = 90) were patients (laypeople) of the university clinic and the remaining half were restorative dentists and prosthodontists with similar levels of clinical experience (at least 3 years of academic training).
Sampling Method: Probability Sample
Enrollment: 180 (Actual)
Dates: Start 2023-06-05 (Actual); Primary Completion 2023-06-12 (Actual); Study Completion 2023-12-22 (Actual)

PRIMARY OUTCOMES:
survey on midline discrepancy at different levels | 10 minutes
  participants was asked to evaluate each image via a Visual analog scale VAS, ranging from point 0 (extremely not esthetic) to point 100 (extremely esthetic).
survey on individual crown width disproportions | 10 minutes
  participants was asked to evaluate each image via a Visual analog scale VAS, ranging from point 0 (extremely not esthetic) to point 100 (extremely esthetic).
survey on distributed crown width disproportions | 10 minutes
  participants was asked to evaluate each image via a Visual analog scale VAS, ranging from point 0 (extremely not esthetic) to point 100 (extremely esthetic).

CONTACTS AND LOCATIONS:
Overall Officials: Bora Korkut, Dr., Principal Investigator — Marmara University Faculty of Dentistry
Locations (1):
- Marmara University Faculty of Dentistry, Istanbul, Turkey (Türkiye)

IPD SHARING:
Plan to Share IPD: Undecided